CLINICAL TRIAL: NCT02772458
Title: Reduced Appetite in Crohn's Disease: Investigating the Role of the Gut Brain Pathways
Brief Title: Reduced Appetite in Crohn's Disease: The Role of the Brain in the Control of Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14038
Record Dates: First submitted 2016-02-11; First posted 2016-05-13 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2017-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; gut brain axis; reduced appetite
MeSH Terms: conditions — Crohn Disease; Anorexia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crohn's Disease (Experimental): Active Crohn's Disease
  Interventions: Other: Dodecanoate acid and saline
- Healthy (Experimental): Healthy volunteers
  Interventions: Other: Dodecanoate acid and saline

INTERVENTIONS:
Other: Dodecanoate acid and saline — Test drink

SUMMARY:
Crohn's disease (CD) is becoming more common, specifically in the western world. One of the main features of this disease is weight loss and malnutrition. Although clinically common, these problems are not well understood. Loss of appetite and symptoms such as tummy aches and bloating are common causes for weight loss in this group of patients. This problem has a strong negative effect on the patients' quality of life and significantly increases the cost of treating CD. Enteroendocrine cells are nutrient sensors in the bowel that relay to the brain to control food intake. Recent evidence has showed that these cells increase in number in active CD and secrete more hormones that negatively affect appetite. The increased levels of these hormones should have an overall negative effect on the brain and thus decrease food intake, bloating, symptoms of sickness. All these symptoms lead to malnutrition. These are hypotheses that require further proof. Current technological advances in magnetic resonance imaging (MRI) has enabled the mapping of changes in activity in important areas in the brain that control food intake. The involvement of the brain in control of food intake is still not fully understood. This work will be the first step in the right direction to start targeting the problems of appetite, weight loss and a poor quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-75 years
2. Ulceration seen at ileocolonoscopy, aiming for a simple endoscopic score for Crohn's disease (SES-CD) of 4-19, in the absence of stricturing disease or,
3. Intestinal inflammation or deep ulceration seen on CT or MR enterography, with the disease activity quantified via the MaRIA score or,
4. Faecal calprotectin of >250µg/g
5. C-Reactive protein >5mg/dl
6. Harvey-Bradshaw index score of 5-16
7. Body mass index (BMI) 18-35
8. As for HV participants, inclusion criteria 1 and 7 will apply.

Exclusion Criteria:

1. Malignant disease
2. BMI <18 and >35
3. Significant cardiovascular or respiratory disease
4. Diabetes mellitus
5. Current Infection
6. Neurological or cognitive impairment; significant physical disability
7. Significant hepatic disease or renal failure
8. Abnormal blood results other than those explained by CD including bleeding diatheses (apart from in the case of HV where all unexplained blood results are an exclusion criteria)
9. Subjects currently participating in (or in the last three months) any other research project
10. pregnancy or breastfeeding or
11. if MRI is contraindicated (e.g. pacemaker).
12. Severe Crohn's disease where a delay in a change in medical treatment for 23 weeks would not be clinically advisable.
13. As for healthy volunteer participants all exclusion criteria apart from no.12.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Changes in Blood Oxygenation Level Dependent (BOLD) response in the brain following a fatty acid test meal in Crohn's patients and healthy controls | 3 years

SECONDARY OUTCOMES:
Changes in arterial spin labeling measures of cerebral blood flow and changes in gut peptide levels following the fatty acid test meal. | 3 years
  The increase or decrease in BOLD signal of the brain following the fatty acid stimuli will be correlated to the gut peptide levels which are listed as follows:
  1. CCK (pmol/ml)
  2. GLP-1 (pM)
  3. PYY (pg/ml)
  4. Ghrelin (ng/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No